CLINICAL TRIAL: NCT06360224
Title: Collect Flow and Ultrasound Images of Coronary Bypass Grafts
Acronym: CASES
Status: Not yet recruiting | Type: Observational
Sponsor: Medistim ASA (Industry)
Responsible Party: Sponsor
Other Study IDs: CASES
Record Dates: First submitted 2024-04-06; First posted 2024-04-11 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Cardiac Bypass Surgery (CABG)

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: MiraQ systems with Transit Time Flow Measurement (TTFM) and High Frequency Ultrasound (HFUS) probes — The objective of this study is to harvest a wide dataset of high quality to allow exploratory analysis and training of machine learning

SUMMARY:
This is a post-market observational, non-interventional, multicenter clinical investigation with the purpose of harvesting high quality data from regular cardiac bypass surgery (CABG).

ELIGIBILITY:
Inclusion Criteria:

* Patient older than 18 years
* Scheduled for CABG
* Understand the nature of the procedure and willingness to comply with the CIP
* Provide written informed consent

Exclusion Criteria:

* Patient younger than 18 years
* Any condition that the investigator believes should exclude participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for cardiac bypass surgery (CABG) that have signed an informed consent form for this study
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-05-15 (Estimated); Primary Completion 2029-05-15 (Estimated); Study Completion 2029-05-15 (Estimated)

PRIMARY OUTCOMES:
Wide and high-quality dataset uploaded to CaseCloud from CABG-procedures. | 1 day

IPD SHARING:
Plan to Share IPD: Undecided